CLINICAL TRIAL: NCT05407935
Title: Early Phase Clinical Trial to Test the Feasibility of an ACT-based Physical Activity Promotion Program for Adults With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34AT011302 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTivity (Experimental): Acceptance and Commitment Therapy for physical activity promotion plus standard physical activity promotion strategies (i.e., goal-setting, self-monitoring)
  Interventions: Behavioral: ACTivity
- Relaxercise (Active Comparator): Relaxation training plus standard physical activity promotion strategies (i.e., goal-setting, self-monitoring)
  Interventions: Behavioral: Relaxercise

INTERVENTIONS:
Behavioral: ACTivity — Acceptance and Commitment Therapy for physical activity promotion plus standard physical activity promotion strategies (i.e., goal-setting, self-monitoring)
  Arms: ACTivity
Behavioral: Relaxercise — Relaxation training plus standard physical activity promotion strategies (i.e., goal-setting, self-monitoring)
  Arms: Relaxercise

SUMMARY:
The goal of the proposed project is to conduct a feasibility clinical trial comparing group-based acceptance and commitment therapy for physical activity, (ACT; ACTivity) to a time- and attention-matched standard PA intervention (i.e., PA education, goal-setting, and self-monitoring) plus relaxation training comparison condition (Relaxercise) among 60 low-active adults (ages 18-65) with elevated depressive symptoms. Participants will be randomized to treatment condition, followed for 6 months, including the 8-week treatment. Participants will be randomized 1:1 to treatment condition, followed for 6 months, including the 8-week treatment, and receive a 6-month YMCA membership to equate access to PA facilities.

ELIGIBILITY:
Inclusion Criteria:

* Elevated depressive symptoms (CES-D score of greater than or equal to 10)
* Low-active (less than 60 minutes per week of moderate intensity PA)
* Willing and able to attend weekly virtual video sessions via Zoom

Exclusion Criteria:

* Regular mindfulness meditation practice (more than once per week)
* Body Mass Index (BMI) less than 18.5 or greater than 40
* History or presence of any condition that may limit or substantially increase the risks of physical activity
* Active suicidal thoughts or behaviors
* Currently participating in any exercise or weight-loss research studies
* Household member is participating in this study
* Does not have a Rhode Island mailing address OR if only Rhode Island mailing address is a PO box
* Unable to receive materials in the mail at residential mailing address
* Does not plan to live in Rhode Island for the next 6 months
* Unable to speak, read, and/or write fluently in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Accelerometry | Baseline, Post-Treatment (8 weeks), 6-months
  Minutes of physical activity weighted by intensity, expressed in metabolic equivalent (MET) minutes per week as determined by accelerometers (Actigraph [model wGT3x-BT]) worn during one-week periods.

SECONDARY OUTCOMES:
Change in Self-report physical activity (Godin) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Self-reported minutes of leisure time physical activity per week weighted by intensity
Change in Self-reported depression symptoms (CES-D) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Score on the Center for Epidemiological Studies Depression Scale (CES-D)

OTHER OUTCOMES:
Change in Physical activity values clarification (valuing questionnaire) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Measures how a person's values align with physical activity
Change in Acceptance of physical activity-related distress (Physical Activity Acceptance Questionnaire) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Measures the extent to which a person can tolerate any distress associated with physical activity
Change in Physical activity-related motivation (Treatment Self-Regulation Questionnaire - Exercise Version) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Measures the extent to which a person is motivated to engage in physical activity
Change in Discomfort intolerance (Discomfort Intolerance Scale) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Measures the extent to which a person can tolerate uncomfortable experiences
Change in Physical activity enjoyment (PACES questionnaire) | Baseline, Mid-Treatment (4 weeks) Post-Treatment (8 weeks), 6-months
  Measures the extent to which a person enjoys physical activity
Change in Credibility and expectancy questionnaire | Week 1 (After the first treatment session)
  Measures perceived credibility and expected benefits of treatment
Change in Client satisfaction questionnaire | Post-Treatment (8 weeks) and following the booster session (12 weeks)
  Measures satisfaction with treatment
Change in Group cohesion questionnaire | Post-Treatment (8 weeks)
  Measures perceived cohesiveness of the treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Da M Wil, Ph.D., Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided